CLINICAL TRIAL: NCT02628236
Title: A Pharmacokinetic Study of Levulan Kerastick (Aminolevulinic Acid HCl) for Topical Solution, 20% Under Maximal Use Conditions
Brief Title: Maximal Use Systemic Exposure Study of Levulan Kerastick (MUSE 2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP0113
Record Dates: First submitted 2015-12-07; First posted 2015-12-11 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Keratosis, Actinic
Keywords: Actinic keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALA (Experimental): 20% aminolevulinic acid applied via Kerastick to individual AK lesions on the upper extremities and covered with occlusive dressing for 3 hours prior to BLU-U treatment
  Interventions: Drug: Aminolevulinic Acid (ALA); Device: BLU-U

INTERVENTIONS:
Drug: Aminolevulinic Acid (ALA) — 20% ALA applied to upper extremities for 3 hours prior to 10 J/cm2 blue light
  Other Names: Levulan Kerastick
Device: BLU-U — 10 J/cm2 of 417 nm blue light delivered at 10 mW/cm2
  Other Names: Blue Light Photodynamic Therapy (PDT)

SUMMARY:
The purpose of this study is to evaluate the potential for systemic exposure of aminolevulinic acid (ALA) and protoporphyrin IX (PpIX) when applied topically under occlusion, in a maximal use setting in patients with multiple actinic keratoses (AK) involving the upper extremities.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 Grade 1/2 AKs on one upper extremity AND
* At least 12 Grade 1/2 AKs on the OTHER upper extremity

Exclusion Criteria:

* Pregnancy
* history of cutaneous photosensitization, porphyria, hypersensitivity to porphyrins or photodermatosis
* lesions suspicious for skin cancer (skin cancer not ruled out by biopsy) or untreated skin cancers within the Treatment Area
* Body Mass Index (BMI) > 32.0 kg/m2
* skin pathology or condition which could interfere with the evaluation of the test product or requires the use of interfering topical or systemic therapy
* significant blood loss within 60 days or donated blood/plasma within 72 hours prior to Visit 2 (Baseline)
* tested positive at screening for human immunodeficiency virus (HIV) or was known to be seropositive for HIV
* a history of lead poisoning or a history of a significant exposure to lead
* tested positive at screening for hepatitis B surface antigen, hepatitis C antibody or had a history of a positive result
* positive drug screen at Screening
* Screening safety labs are clinically significant in the opinion of the investigator
* major surgery within 30 days prior to Visit 2 (Baseline) or plans to have surgery during the study
* Subject is immunosuppressed
* currently enrolled in an investigational drug or device study
* has received an investigational drug or been treated with an investigational device within 30 days prior to Visit 2 (Baseline)
* known sensitivity to one or more of the vehicle components (ethyl alcohol, isopropyl alcohol, laureth 4, polyethylene glycol)
* use of the following topical preparations on the extremities to be treated:

  * Keratolytics including urea (greater than 5%), alpha hydroxyacids [e.g.glycolic acid, lactic acid, etc. greater than 5%], salicylic acid (greater than 2%) within 2 days of initiation of treatment
  * Cryotherapy within 2 weeks of initiation of treatment
  * Retinoids, including tazarotene, adapalene, tretinoin, retinol, within 4 weeks of initiation of treatment
  * Microdermabrasion, laser ablative treatments, ALA-PDT, chemical peels, 5-FU, diclofenac, imiquimod or other topical treatments for AK within 8 weeks of initiation of treatment
* use of systemic retinoid therapy within 6 months of initiation of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Marcus, MD, PhD, Study Director — DUSA Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - DermResearch, Inc., Austin, Texas
  - J&J Studies, Inc, College Station, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ALA-PDT: 20% aminolevulinic acid applied via Kerastick to individual AK lesions on the upper extremities and covered with occlusive dressing for 3 hours prior to BLU-U treatment
  Aminolevulinic Acid (ALA): 20% ALA applied to upper extremities for 3 hours prior to 10 J/cm2 blue light
  BLU-U: 10 J/cm2 of 417 nm blue light delivered at 10 mW/cm2
Period: Overall Study
Arm/Group | ALA-PDT
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Maximum Baseline Corrected Plasma Concentration (Cmax) for ALA
Description: Maximum baseline corrected plasma concentration (Cmax) for ALA over the 24 hour sampling time period. Blood samples were taken before ALA application and at 15 and 30 minutes, 1, 2, 4, 8, 12, 16, 24, 36 and 48 hours following study medication application.
Time Frame: 2 days
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
ng/mL | 39.05 (319.7)

2. Primary Outcome: Time at Which Cmax is Attained (Tmax) for ALA
Description: Time of the maximum baseline corrected plasma concentration for ALA measured at at 15 and 30 minutes, 1, 2, 4, 8, 12, 16, 24, 36 and 48 hours following study medication application.If a maximum value occurred at more than one timepoint Tmax is defined as the first timepoint with this value.
Time Frame: 2 days
Measure: Median (Full Range); unit: hours
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
hours | 2 [0.25 to 36]

3. Primary Outcome: AUCt
Description: AUCt is the area under the baseline corrected plasma concentration-time profile up to the last quantifiable/non-negative plasma concentration
Time Frame: 0, 15, 30 minutes, and 1, 2, 4, 8, 12, 16, 24 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
ng*hr/mL | 182.1 (111.6)

4. Primary Outcome: The Terminal Exponential Half-life (T1/2,z) for ALA
Description: The terminal slope was calculated by linear least squares regression of the log plasma concentration-time data. The terminal exponential half-life (T1/2,z) will be calculated as 0.693 divided by the absolute value of slope.
Time Frame: 2 days
Population: T1/2,z could not be determined in 11 subjects
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | ALA-PDT
Number analyzed (Participants) | 3
hours | 5.386 (253.7)

5. Primary Outcome: Maximum Baseline Corrected Plasma Concentration (Cmax) for PpIX
Description: Maximum baseline corrected plasma concentration (Cmax) for PpIX over the 48 hour sampling time period. Blood samples were taken before ALA application and at 15 and 30 minutes, 1, 2, 4, 8, 12, 16, 24, 36 and 48 hours following study medication application.
Time Frame: 2 days
Population: For 50% of the subjects, more than 50% of the PpIX plasma concentrations following topical application of ALA HCI were less than the predose plasma concentration. Therefore, negative values were set to 0 to evaluate median baseline corrected plasma concentration.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
ng/mL | 0.735 [0 to 2.3]

6. Primary Outcome: Time at Which Cmax is Attained (Tmax) for PpIX
Description: Time of the maximum baseline corrected plasma concentration for PpIX measured at at 15 and 30 minutes, 1, 2, 4, 8, 12, 16, 24, 36 and 48 hours following study medication application.If a maximum value occurred at more than one timepoint Tmax is defined as the first timepoint with this value.
Time Frame: 2 days
Population: One subject had tmax that could not be determined.
Measure: Median (Full Range); unit: hours
Arm/Group | ALA-PDT
Number analyzed (Participants) | 13
hours | 12 [0.25 to 48]

7. Primary Outcome: AUCBL for PpIX
Description: The area under the concentration time-curve assuming the baseline observed plasma concentration existed from time 0 to tlast.
Time Frame: 0, 15, 30 minutes, and 1, 2, 4, 8, 12, 16, 24, 36 and 48 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
ng*hr/mL | 77.34 (98.04)

8. Primary Outcome: AUCt for PpIX
Description: The area under the observed plasma concentration time-curve from time 0 to the last quantifiable plasma concentration.
Time Frame: 0, 15, 30 minutes, and 1, 2, 4, 8, 12, 16, 24, 36 and 48 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
ng*hr/mL | 77.00 (59.16)

9. Primary Outcome: AUCt/AUCBL for PpIX
Description: The ratio of AUCt to AUCBL for PpIX
Time Frame: 0, 15, 30 minutes, and 1, 2, 4, 8, 12, 16, 24, 36 and 48 hours post-dose
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
ratio | 0.9956 [0.831 to 1.19]

10. Secondary Outcome: Hyperpigmentation
Description: HYPERPIGMENTATION SCALE Grade 0 = No hyperpigmentation Grade 1 = Light hyperpigmentation involving small areas Grade 2 = Moderate hyperpigmentation involving small areas; light hyperpigmentation involving moderate areas Grade 3 = Moderate hyperpigmentation involving moderate sized areas; light hyperpigmentation involving large areas; small areas of marked hyperpigmentation Grade 4 = Marked hyperpigmentation involving moderate or large sized areas
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 6
  Grade 1 | 7
  Grade 2 | 1
  Grade 3 | 0
  Grade 4 | 0

11. Secondary Outcome: Hyperpigmentation
Description: as for outcome 10
Time Frame: 24 hours after PDT
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 7
  Grade 1 | 6
  Grade 2 | 1
  Grade 3 | 0
  Grade 4 | 0

12. Secondary Outcome: Hyperpigmentation
Description: as for outcome 10
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 7
  Grade 1 | 6
  Grade 2 | 1
  Grade 3 | 0
  Grade 4 | 0

13. Secondary Outcome: Hypopigmentation
Description: HYPOPIGMENTATION SCALE Grade 0 = No hypopigmentation Grade 1 = Light hypopigmentation involving small areas Grade 2 = Moderate hypopigmentation involving small areas; light hypopigmentation involving moderate areas Grade 3 = Moderate hypopigmentation involving moderate sized areas; light hypopigmentation involving large areas; small areas of marked hypopigmentation Grade 4 = Marked hypopigmentation involving moderate or large sized areas
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 8
  Grade 1 | 6
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

14. Secondary Outcome: Hypopigmentation
Description: as for outcome 13
Time Frame: 24 hours after PDT
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 8
  Grade 1 | 6
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

15. Secondary Outcome: Hypopigmentation
Description: as for outcome 13
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 8
  Grade 1 | 6
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

16. Secondary Outcome: Erythema
Description: Erythema Scale - Grade 0 = None Grade 1 = Minimal - barely perceptible erythema Grade 2 = Mild - predominantly minimal erythema (pink) in the treated area with or without a few isolated areas of more intense erythema Grade 3 = Moderate - predominantly moderate erythema (red) in the treated area with or without a few isolated areas of intense erythema (bright red) Grade 4 = Severe - predominantly intense erythema (bright red) in the treated area with or without a few isolated areas of very intense (fiery red) erythema
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 11
  Grade 1 | 1
  Grade 2 | 2
  Grade 3 | 0
  Grade 4 | 0

17. Secondary Outcome: Erythema
Description: as for outcome 16
Time Frame: 5 Minutes after PDT
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 4
  Grade 1 | 2
  Grade 2 | 5
  Grade 3 | 3
  Grade 4 | 0

18. Secondary Outcome: Erythema
Description: as for outcome 16
Time Frame: 24 hours after PDT
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 0
  Grade 1 | 3
  Grade 2 | 4
  Grade 3 | 7
  Grade 4 | 0

19. Secondary Outcome: Erythema
Description: as for outcome 16
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 7
  Grade 1 | 6
  Grade 2 | 1
  Grade 3 | 0
  Grade 4 | 0

20. Secondary Outcome: Edema
Description: EDEMA SCALE Grade 0 = None Grade 1 = Minimal - scant, rare edema Grade 2 = Mild - easily seen edema, minimally palpable, involving up to 1/3 of the treatment area Grade 3 = Moderate - easily seen edema and typically palpable, involving between 1/3 to 2/3 of the treatment area Grade 4 = Severe - easily seen edema, indurated in some areas, involving over 2/3 of the treatment area
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 14
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

21. Secondary Outcome: Edema
Description: as for outcome 20
Time Frame: 5 Minutes after PDT
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 8
  Grade 1 | 5
  Grade 2 | 1
  Grade 3 | 0
  Grade 4 | 0

22. Secondary Outcome: Edema
Description: as for outcome 20
Time Frame: 24 hours after PDT
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 8
  Grade 1 | 3
  Grade 2 | 3
  Grade 3 | 0
  Grade 4 | 0

23. Secondary Outcome: Edema
Description: as for outcome 20
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 14
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

24. Secondary Outcome: Stinging/Burning
Description: STINGING AND BURNING SCALE Grade 0 = None Grade 1 = Minimal, barely perceptible -tolerable and little discomfort Grade 2 = Moderate - tolerable, but causes some discomfort Grade 3 = Severe - very uncomfortable or intolerable
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 13
  Grade 1 | 1
  Grade 2 | 0
  Grade 3 | 0

25. Secondary Outcome: Stinging/Burning
Description: as for outcome 24
Time Frame: Intraprocedure
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 0
  Grade 1 | 6
  Grade 2 | 8
  Grade 3 | 0

26. Secondary Outcome: Stinging/Burning
Description: as for outcome 24
Time Frame: 5 Minutes after photodynamic therapy
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 6
  Grade 1 | 5
  Grade 2 | 3
  Grade 3 | 0

27. Secondary Outcome: Stinging/Burning
Description: as for outcome 24
Time Frame: 24 hours after PDT
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  g | 10
  Grade 1 | 4
  Grade 2 | 0
  Grade 3 | 0

28. Secondary Outcome: Stinging/Burning
Description: as for outcome 24
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 13
  Grade 1 | 1
  Grade 2 | 0
  Grade 3 | 0

29. Secondary Outcome: Scaling and Dryness
Description: SCALING AND DRYNESS SCALE Grade 0 = None Grade 1 = Minimal - barely perceptible desquamation Grade 2 = Mild - limited areas of fine desquamation in up to 1/3 of the treatment area Grade 3 = Moderate - fine desquamation involving 1/3 to 2/3 of the treatment area or limited areas of coarser scaling Grade 4 = Severe - coarser scaling involving more than 2/3 of the treatment area or limited areas of very coarse scaling
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 12
  Grade 1 | 2
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

30. Secondary Outcome: Scaling and Dryness at Visit 4
Description: as for outcome 29
Time Frame: 24 hours after PDT
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 9
  Grade 1 | 3
  Grade 2 | 1
  Grade 3 | 1
  Grade 4 | 0

31. Secondary Outcome: Scaling and Dryness
Description: as for outcome 29
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 9
  Grade 1 | 5
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

32. Secondary Outcome: OOZING/VESICULATION/CRUSTING
Description: OOZING/VESICULATION/CRUSTING Grade 0 = None Grade 1 = Minimal - a single area of oozing, vesiculation or crusting 3 mm diameter or less in size Grade 2 = Mild - two to four areas of oozing, vesiculation or crusting 3 mm diameter or less in size OR a single area larger than 3 mm diameter in size Grade 3 = Moderate - more than a single area of oozing, vesiculation or crusting larger than 3 mm diameter in size or more than four areas of 3 mm diameter or less in size Grade 4 = Severe - any degree of oozing, vesiculation or crusting greater than (3) above
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 14
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

33. Secondary Outcome: OOZING/VESICULATION/CRUSTING
Description: as for outcome 32
Time Frame: 24 hours after PDT
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 13
  Grade 1 | 1
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

34. Secondary Outcome: OOZING/VESICULATION/CRUSTING
Description: as for outcome 32
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | ALA-PDT
Number analyzed (Participants) | 14
Participants
  Grade 0 | 14
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | ALA-PDT
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALA-PDT (N=14)
deep vein thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
First publication of results will be made by the Sponsor. If publication is not submitted within 12 months after the date of study final report, the PI may publish the results from the site individually, subject to compliance with the other terms of the clinical trial agreement, including a requirement that the PI provide a draft of the publication for the sponsor's review 30 days before submission for publication so that sponsor can review the publication for confidential information